CLINICAL TRIAL: NCT02425085
Title: Comparative Study of Multi-endodiathermy Retinectomy Versus Relaxing Retinectomy for Retinal Re-detachment in Silicone Oil Filled Eye
Brief Title: Comparative Study of Multi-endodiathermy Retinectomy Versus Relaxing Retinectomy for Retinal Re-detachment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiaofeng Lin, vice-president, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MER201504
Record Dates: First submitted 2015-04-16; First posted 2015-04-23 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Retinal Redetachment in Silicone Oil-filled Eyes
Keywords: retinectomy; endodiathermy; inferior; retinal redetachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- multi-endodiathermy retinectomy group (Experimental): Patients receive multi-endodiathermy retinectomy
  Interventions: Procedure: multi-endodiathermy retinectomy
- relaxing retinectomy (Active Comparator): Patients receive relaxing retinectomy
  Interventions: Procedure: relaxing retinectomy

INTERVENTIONS:
Procedure: multi-endodiathermy retinectomy — patients will receive multi-endodiathermy retinectomy; 6 months later, patients will receive the removal of intraocular silicone oil.
  Arms: multi-endodiathermy retinectomy group
Procedure: relaxing retinectomy — patients will receive relaxing retinectomy; 6 months later, patients will receive the removal of intraocular silicone oil.
  Arms: relaxing retinectomy

SUMMARY:
Previous pilot study has demonstrated that the novel multi-endodiathermy retinectomy is feasible, effective and safe for inferior retinal redetachments in the silicone oil-filled eyes of adults over a 3-month observation.

Here, the investigators conduct this randomized and multicenter clinical trial to compare the efficacy and safety between multi-endodiathermy retinectomy and relaxing retinectomy.

DETAILED DESCRIPTION:
The relaxing retinectomy is a useful surgery for retinal re-detachment in eyes with silicone oil filled. However, it has some obvious disadvantages such as the cut of the normal retina surrounding, leaving a large area of retinal deficiency and significant exposure of retinal pigment epithelium and choroid membranes.

We proposed a novel multi-endodiathermy retinectomy as a potential surgery. A pilot study has demonstrated that the novel multi-endodiathermy retinectomy is feasible, effective and safe for inferior retinal redetachments in the silicone oil-filled eyes of adults over a 3-month observation.

Here, the investigators conduct this randomized and multicenter clinical trial to compare the efficacy and safety between multi-endodiathermy retinectomy and relaxing retinectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years, male or female;
* The primary retinal detachment was caused by ocular trauma, and the vitreous body is filled with silicone oil now;
* The presence of inferior retinal re-detachment located among 3-9 o'clock.

Exclusion Criteria:

* Location of the re-detached retina is not mainly in the inferior of the eye;
* The fundus is unobservable because of severe corneal opacity;
* The contralateral eye is non-functional;
* Serious heart, lung, liver and kidney dysfunction.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 328 (Estimated)
Dates: Start 2015-04; Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
retinal reattachment | 3 months after retinectomy

SECONDARY OUTCOMES:
operative duration | from the end of former silicone oil removal to the end of the new silicone oil fill
visual acuity | 1 day before surgery; 3 days, 1 week, 2 weeks, 4 weeks and 3 months after retinectomy; 3 days, 1 week, 2 weeks, 4 weeks and 3 months after silicone oil removal.
intraocular pressure | 1 day before surgery; 3 days, 1 week, 2 weeks, 4 weeks and 3 months after retinectomy; 3 days, 1 week, 2 weeks, 4 weeks and 3 months after silicone oil removal.
the incidence of intraocular hemorrhage | during retinectomy
degree of recurrent PVR | 1 day before surgery; 3 days, 1 week, 2 weeks, 4 weeks and 3 months after retinectomy; 3 days, 1 week, 2 weeks, 4 weeks and 3 months after silicone oil removal.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Lin, M.D, Principal Investigator — Zhongshan Ophthalmic Center of Sun yat-sen Universtiy
Locations (3):
- China (3):
  - Zhongshan Ophthalmic Center of Sun yat-sen Universtiy, Guangzhou, Guangdong
  - Shenzhen Ophthalmic Center, Shenzhen, Guangdong
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

REFERENCES:
- [Background] Romaniuk VM. Ocular trauma and other catastrophes. Emerg Med Clin North Am. 2013 May;31(2):399-411. doi: 10.1016/j.emc.2013.02.003. PMID 23601479
- [Background] Han DP, Lewis MT, Kuhn EM, Abrams GW, Mieler WF, Williams GA, Aaberg TM. Relaxing retinotomies and retinectomies. Surgical results and predictors of visual outcome. Arch Ophthalmol. 1990 May;108(5):694-7. doi: 10.1001/archopht.1990.01070070080039. PMID 2334327
- [Background] Kolomeyer AM, Grigorian RA, Mostafavi D, Bhagat N, Zarbin MA. 360 degrees retinectomy for the treatment of complex retinal detachment. Retina. 2011 Feb;31(2):266-74. doi: 10.1097/IAE.0b013e3181eef2c7. PMID 21124255
- [Background] Machemer R. [Cutting of the retina: a means of therapy for retinal reattachment (author's transl)]. Klin Monbl Augenheilkd. 1979 Nov;175(5):597-601. German. PMID 547089